CLINICAL TRIAL: NCT05212402
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Physiological, Biochemical, and Psychometric Impacts of a Brand-Specific Hemp-Derived Cannabidiol Product in Healthy Adults
Brief Title: Assessing the Effects of a Cannabidiol Derived From Hemp Supplement in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00115662
Record Dates: First submitted 2021-12-06; First posted 2022-01-28 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Healthy; Safety Issues
MeSH Terms: interventions — Cannabinol

STUDY DESIGN:
Intervention Model Description: Between subjects study design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded of the subjects and research staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): 28 participants will be given the test product (TP)
  Interventions: Dietary Supplement: Cannabinol
- Placebo (Placebo Comparator): 28 participants will be given the placebo product.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cannabinol — Prospective,1:1 randomization and stratified by birth sex, and double-blinded to the condition of subjects.
  Arms: Test Product
Other: Placebo — Prospective,1:1 randomization and stratified by birth sex, and double-blinded to the condition of subjects.
  Arms: Placebo

SUMMARY:
The purpose of this prospective, randomized, double-blind, placebo-controlled trial is to assess the physiological, biochemical, and psychometric impacts of a brand-specific hemp-derived cannabidiol product in a sample of healthy adults.

DETAILED DESCRIPTION:
Cannabis contains several phyto-cannabinoids among which Δ9-tetrahydrocannabinol (THC) and cannabidiol (CBD) are most widely known. THC is the main compound responsible for the psychoactive properties and also deemed responsible for several side-effects associated with cannabis. CBD, on the other hand, is not a strong cannabinoid receptor agonist and lacks psychotropic activity. However, due to its affinity for several other target sites, it is being studied for potential pharmacological properties. The diverse range of interactions at different receptor sites in the human body is believed to be responsible for therapeutic efficacy of CBD in treating kidney fibrosis, metabolic syndrome, anorexia, obesity, amelioration of osteoarthritis as well as several other musculoskeletal diseases. Recent research has also explored the use of CBD to relieve stress and depression, likely due to its agonistic influence on the 5-HT3 receptors as well as improving hippocampal neural growth and development. CBD has also been studied for its anti-oxidant activity, deemed on-par to that of Vitamin C in laboratory studies. The effect of CBD on inflammation and the immune system has been studied. The sedative effects of CBD have been investigated for the potential use of CBD as an anxiolytic and to improve mood as well as sleep. Recent studies have also explored the analgesic and pain-relieving properties of CBD, making it a suitable candidate that needs further investigations. Interestingly, a recent systematic review explored the use of CBD in viral diseases, with several pre-clinical studies indicating CBD as an effective candidate against viral disease. With the spread of the coronavirus disease (COVID-19) pandemic, there has been a strong interest in developing therapies to eliminate or reduce the risk of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. SARS-CoV-2 uses Angiotensin Converting Enzyme (ACE) receptors to gain entry into the human body and penetrate the respiratory system. In a recent in vitro study, pretreatment with CBD in cells expressing ACE-2 receptor was effective in inhibiting the replication of SARS-CoV-2 in those cells. This is an interesting finding where further research is needed to study the influence of CBD consumption on ACE activity. Several studies of CBD safety have demonstrated lack of any safety concerns over a range of different doses. A recent safety study of CBD by Bergamaschi et al. demonstrated absence of any influence on the central nervous system, vital signs or mood changes as well as lack of any side effect observed for doses up to 1500 mg/day (orally) or 30 mg/day (intravenously).It has been hypothesized that the trace amounts of THC present within the CBD extract could potentially be responsible for any side-effects. Therefore, CBD is considered very safe for human consumption in the dose being tested in this study (<200mg/day). Additional clinical research is required to confirm and support therapeutic use of CBD for being effective in modulating ACE expression, mood, stress, anti-inflammatory, antioxidant, immunomodulating, sedative & anxiolytic, analgesic, pain relieving and anti-viral therapeutic claims. This research will also help to understand any safety issues with the long-term regular use of CBD on healthy adults. Therefore, this prospective, randomized, double-blind, placebo controlled study will be conducted to explore the physiologic, biochemical, and psychometric impacts of a brand-specific hemp-derived CBD product in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* body mass index of 19.0 to 34.9 kg/m2 (normal weight through Class I obesity)
* Agree to refrain from alcohol consumption for at least 48 hours prior to each visit.
* Willing to practice acceptable measures of birth control and sexually transmitted infections prevention by using double-barrier contraceptive measures (both males and females) throughout the study duration.
* Willing and able to agree to the requirements and restrictions of this study including fasting before blood draw on all visits for laboratory assessment.
* Willing to give voluntary consent, be able to understand and read the questionnaires, carry out all study-related procedures, communicate effectively with the study staff, and agree to allow any study related evaluations.

Exclusion Criteria:

* Have a known sensitivity or allergy to any of the investigational products or their ingredients.
* Female participants who are lactating, pregnant or planning to become pregnant during the study as confirmed at the baseline (visit 2) or male participants of reproductive potential in a heterosexual relationship planning a pregnancy as confirmed at the baseline visit.
* Documented medical history of immune disorder (such as Human immunodeficiency Virus/Acquired immunodeficiency syndrome), hepatitis B or hepatitis C, or reported immune disorder diagnosis.
* Active psychiatric disorder requiring hospitalization within the 12 months prior to screening or currently on medication(s) to treat any psychiatric disorder(s).
* Any cognitive impairment that would, in the opinion of the Investigator, preclude study participation or compliance with study procedures (e.g., Alzheimer's, dementia).
* History of malignancy or those with any first-degree relatives with a history of cancer (e.g., familial cancer disorders) within 5 years.
* History of clinically significant cardiovascular, respiratory, renal, cerebrovascular, metabolic, pulmonary, gastrointestinal, neurological, hematological, autoimmune, lymphatic, psychiatric, chronic pain and sleep disorders, hepatobiliary (with the exception of Gilbert's syndrome or asymptomatic gallstones) or endocrine disorders, including individuals with Type I or Type II diabetes, or other clinically significant medical condition that, in the opinion of the Investigator, may preclude safe study participation.
* Participants with controlled or uncontrolled hypertension including stage 1 hypertension (systolic blood pressure ≥129 mmHg and diastolic blood pressure ≥89 mmHg).
* Participants who are on medications as prescribed for any of the aforementioned exclusionary criteria. Participants on stable dose of thyroid medication (no dosage changes within last 3 months) are acceptable.
* Consumption of prescription or non-prescription: angiotensin converting enzyme inhibitors, angiotensin receptor blockers, barbiturates, cocaine, ethanol, selective serotonin reuptake inhibitor, protease inhibitors, warfarin, sildenafil, theophylline, tricyclic antidepressants and any other medications
* Receipt or use of an investigational product in another research study within 30 days or 5 half lives (whichever is longer) prior to baseline (visit 2) or currently participating in another study
* Receipt or use of an investigational product in another research study within 30 days or 5 half lives (whichever is longer) prior to baseline (visit 2) or currently participating in another study
* Current or recent use (within one month prior to visit 2) of cannabis (e.g., marijuana) or cannabis related products (e.g., CBD) in any ingestible or inhalable forms.
* Positive urine drug test for THC or drugs of abuse (Amphetamine, cocaine, marijuana, methamphetamine, and opiates) at baseline (visit 2).
* Safety blood tests at screening more than 2 times the upper limit of normal (ULN) for liver or kidney function tests.
* Safety blood tests at screening more than 2 times the upper limit of normal (ULN) for liver or kidney function tests.
* Fasting blood glucose of ≥160 mg/dL (after a repeat that confirms the original result) at screening.
* Any other condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in angiotensin-renin converting enzyme (ACE) | Baseline, Month 1, Month 2, Month 3
  To determine if the test product (TP) has any effect on the activity of angiotensin-renin converting enzyme (ACE) compared to placebo
Changes in white blood cell count | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on white blood cell count compared to placebo
Changes in red blood cell count | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on red blood cell count compared to placebo
Changes in hemoglobin | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on hemoglobin compared to placebo
Changes in hematocrit | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on hematocrit compared to placebo
Changes in mean corpuscular volume | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on mean corpuscular volume compared to placebo
Changes in mean corpuscular hemoglobin concentration | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on mean corpuscular hemoglobin concentration compared to placebo
Changes in red blood cell distribution width | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on red blood cell distribution width concentration compared to placebo
Changes in platelet count | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on platelet count compared to placebo
Changes in mean platelet volume | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on mean platelet volume compared to placebo
Changes in absolute and relative neutrophils | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on absolute and relative neutrophils compared to placebo
Changes in absolute and relative lymphocytes | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on absolute and relative lymphocytes compared to placebo
Changes in absolute and relative monocytes | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on absolute and relative monocytes compared to placebo
Changes in absolute and relative eosinophils | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on absolute and relative eosinophils compared to placebo
Changes in absolute and relative basophils | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on absolute and relative basophils compared to placebo
Changes in TNF-alpha | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on TNF-alpha compared to placebo
Changes in interleukin-6 | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on interleukin-6 compared to placebo
Changes in interleukin-10 | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on interleukin-10 compared to placebo
Changes in cold and flu prevalence | Baseline, Month 3
  To determine if the TP has an impact on number of days of lost productivity (days taken off from work or school) due to cold/flu symptoms compared to placebo
Changes in subjective stress levels | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on stress levels assessed by Cohen's perceived stress scale compared to placebo. The minimum value is 0 and the maximum value is 40. Higher scores mean a worse outcome.
Changes in sleep quality | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on sleep quality assessed by Pittsburgh Sleep Quality Index compared to placebo. The minimum score is 0 and the maximum score is 40. Higher scores mean a worse outcome.
Changes in total mood disturbances | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on total mood disturbance assessed by the Profile of Mood States (POMS) compared to placebo The total mood is calculated by adding the negative subscales (tension, depression, fatigue, confusion, and anger) subtracting the positive subscales (vigor, esteem-related affect).
Changes in fatigue-inertia | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on fatigue-inertia (POMS sub-score) compared to placebo. Min 0, Max 28, higher scores may be associated with worse outcomes.
Changes in anger-hostility | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on anger-hostility (POMS sub-score) compared to placebo. Min 0, max 48, higher scores are associated with worse outcomes.
Changes in vigor-activity | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on vigor-activity (POMS sub-score) compared to placebo. Min 0, max 32, higher scores are associated with better outcomes.
Changes in confusion-bewilderment | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on confusion-bewilderment (POMS sub-score) compared to placebo. Min 0, max 28, and higher scores are associated with worse outcomes.
Changes in depression-dejection | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on depression-dejection (POMS sub-score) compared to placebo. Min 0, max 60, and higher scores are associated with worse outcomes.
Changes in tension-anxiety | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on tension-anxiety (POMS sub-score) compared to placebo. Min 0, max 60, higher scores are associated with worse outcomes.
Changes in Overall Body Pain/Discomfort Scale | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on body pain and discomfort assessed by the Overall Body Pain/Discomfort Scale compared to placebo, which is a validated dually anchored Likert 10-point scale. Min value is 0, the max is 10, and a higher value is a worse outcome.
Changes in foundation pain | Baseline, Month 1, Month 2, Month 3
  To determine if the TP has an impact on foundation pain index which is calculated from urinalysis compared to placebo. Min 0 and Max 100, higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Changes in AST as a marker of liver function | Baseline, Month 3
  To determine if the TP has an impact on serum AST as a marker of liver function assessed using a comprehensive metabolic panel compared to placebo
Changes in ALT as a marker of liver function | Baseline, Month 3
  To determine if the TP has an impact on serum ALT as a marker of liver function assessed using a comprehensive metabolic panel compared to placebo
Changes in alkaline phosphatase as a marker of liver function | Baseline, Month 3
  To determine if the TP has an impact on serum alkaline phosphatase as a marker of liver function assessed using a comprehensive metabolic panel compared to placebo
Changes in creatinine as a marker of kidney function | Baseline, Month 3
  To determine if the TP has an impact on creatinine as a marker of kidney function assessed using a comprehensive metabolic panel compared to placebo
Changes in potassium as a marker of kidney function | Baseline, Month 3
  To determine if the TP has an impact on potassium as a marker of kidney function assessed using a comprehensive metabolic panel compared to placebo
Changes in blood urea nitrogen as a marker of kidney function | Baseline, Month 3
  To determine if the TP has an impact on blood urea nitrogen as a marker of kidney function assessed using a comprehensive metabolic panel compared to placebo
Changes in blood glucose | Baseline, Month 3
  To determine if the TP has an impact on blood glucose assessed using a comprehensive metabolic panel compared to placebo
Changes in electrolyte balance | Baseline, Month 3
  To determine if the TP has an impact on electrolyte balance assessed using a comprehensive metabolic panel compared to placebo
Changes in serum albumin | Baseline, Month 3
  To determine if the TP has an impact on serum albumin assessed using a comprehensive metabolic panel compared to placebo
Changes in serum albumin/globulin ratio | Baseline, Month 3
  To determine if the TP has an impact on serum albumin/globulin ratio assessed using a comprehensive metabolic panel compared to placebo
Changes in total serum bilirubin serum | Baseline, Month 3
  To determine if the TP has an impact on total bilirubin assessed using a comprehensive metabolic panel compared to placebo
Changes in total serum protein | Baseline, Month 3
  To determine if the TP has an impact on total serum protein assessed using a comprehensive metabolic panel compared to placebo
Changes in blood urea nitrogen | Baseline, Month 3
  To determine if the TP has an impact on blood urea nitrogen assessed using a comprehensive metabolic panel compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No